CLINICAL TRIAL: NCT01937507
Title: Pilot Study of Hepatic Arterial Infusion (HAI) With Oxaliplatin, Folinic Acid and 5 Fluorouracil (FOLFOX) in Heavily Pre-Treated Patients With Liver-Predominant Metastasis From Breast Cancer
Brief Title: Hepatic Artery Infusion With FOLFOX in Liver Metastasis From Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Decision
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-20
Record Dates: First submitted 2013-06-24; First posted 2013-09-09 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HAI with FOLFOX (Experimental): Hepatic Artery Infusion with Oxaliplatin, 5FU, and Folinic Acid
  Interventions: Drug: HAI with FOLFOX

INTERVENTIONS:
Drug: HAI with FOLFOX — HAI with FOLFOX q 3 weeks
  Other Names: Hepatic Artery Infusion

SUMMARY:
Deliver oxliplatin and 5-FU via HAI to breast cancer patients with liver-only or liver-predominant metastases who have failed at least one line of systemic chemotherapy in metastatic setting.

DETAILED DESCRIPTION:
In this pilot study, the investigators will deliver oxliplatin and 5-FU via HAI to breast cancer patients with liver-only or liver-predominant metastases who have failed at least one line of systemic chemotherapy in metastatic setting. The investigators hypothesize that HAI chemotherapy will be able to convert some patients to surgical resection candidates, or/and to overcome chemo-resistance of liver metastases to systemic i.v. chemotherapy for some clinically fit, heavily pre-treated patients.

ELIGIBILITY:
Inclusion Criteria:

1. Performance status ECOG 0-2 and a life expectancy of >3 months.
2. Patients were required to have measurable disease in the liver, defined as lesions measuring >1 cm in largest diameter on spiral-computed tomography (CT) or magnetic resonance imaging (MRI)
3. Histologically confirmed metastatic advanced solid tumors involving the liver, liver replacement less than 70%
4. No bevacizumab (avastin) use within 4 weeks prior to enrollment.
5. Absence of portal vein thrombosis
6. Not a surgical candidate or patients refuge surgery at the time of enrollment
7. Loss of response to at least 1 line of systemic chemotherapy in metastatic setting
8. An asymptomatic extra-hepatic disease is allowed, provided that the extent of the metastatic disease in the liver represented the bulk of the metastatic disease.
9. History of liver-directed therapy is eligible at the investigator's discretion.
10. Adequate renal function with a calculated creatinine clearance greater than 60 mL/min.
11. Hepatic function as follows: Total Bilirubin ≤3 mg/dL, AST ≤5 times upper normal reference value, or ALT ≤ 5 times upper normal reference value.
12. Adequate bone marrow function (ANC ≥1500 cells/uL; PLT ≥ 100,000 cells/uL) before each therapy.
13. At least three weeks from previous immunotherapy, chemotherapy or radiotherapy before being enrolled in this study.
14. All females in childbearing age MUST have a negative serum HCG test unless patients have prior hysterectomy.

Exclusion Criteria:

1. Clinical or radiographic evidence of moderate amount of ascites.
2. History of cirrhosis with Child-Pugh class B or C.
3. Pregnant or lactating females.
4. Inability to complete informed consent process and adhere to protocol treatment plan and follow-up requirements.
5. Patients receiving any other investigational agents.
6. Patients with bleeding diathesis (clinical bleeding, prothrombin time =/> 1.5 X upper institutional normal value, INR =/> 1.5, activated partial thromboplastin time aPTT =/> 1.5 X upper institutional normal value), active gastric or duodenal ulcer.
7. History of thrombophilia, recurrent DVTs, diagnosis of phospholipid syndrome.
8. Past or current history of malignancy other than breast cancer with the exception of treated non-melanoma skin cancer or carcinoma in situ of the cervix, or other cancers cured by local therapy alone and a DFS ≥5 years.
9. Concurrent severe illness such as active infection, or psychiatric illness/social situations that would limit safety and compliance with study requirements.
10. Patients with clinically significant cardiovascular disease: myocardial infarction or unstable angina within 6 months, New York Heart Association Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, unstable angina pectoris, clinically significant peripheral vascular disease
11. Patients have untreated brain metastasis requiring or leptomeningeal metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiaxin Niu, MD, Principal Investigator — Western Regional Medical Center
Locations (1):
- Western Regional Medical Center Inc, Goodyear, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HAI With FOLFOX
Started | 2
Completed | 0
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | HAI With FOLFOX
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Determine Response Rate (RR) of HAI With Oxaliplatin/5-FU Every Three Weeks in Heavily Pre-treated Patients With Advanced Breast Cancer With Metastasis to the Liver.
Description: To determine response rate (RR) of HAI with oxaliplatin/5-FU every three weeks in heavily pre-treated patients with advanced breast cancer with metastasis to the liver.
Time Frame: One year
Population: Data was not collected
Arm/Group | HAI With FOLFOX
Number analyzed (Participants) | 0

2. Primary Outcome: Determine Time to Intra-hepatic Progression (TIP) of HAI With Oxaliplatin/5-FU Every Three Weeks in Heavily Pre-treated Patients With Advanced Breast Cancer With Metastasis to the Liver.
Description: To determine time to intra-hepatic progression (TIP) of HAI with oxaliplatin/5-FU every three weeks in heavily pre-treated patients with advanced breast cancer with metastasis to the liver.
Time Frame: One year
Population: Data was not collected
Arm/Group | HAI With FOLFOX
Number analyzed (Participants) | 0

3. Primary Outcome: Extra-hepatic Progression (TEP) of HAI With Oxaliplatin/5-FU
Description: To determine time to extra-hepatic progression (TEP) of HAI with oxaliplatin/5-FU every three weeks in heavily pre-treated patients with advanced breast cancer with metastasis to the liver.
Time Frame: One year
Population: Data was not collected
Arm/Group | HAI With FOLFOX
Number analyzed (Participants) | 0

4. Secondary Outcome: To Document the Toxicity, Tolerability of the Therapy in This Population.
Description: Document the toxicity and tolerability of the therapy using the following CBC with differential, BUN, creatinine, liver function tests,CA 15-3, CA 27.29, Circulating tumor cells (CTCs)and Restaging radiographic studies (MRI or CT liver protocol).
Time Frame: one year
Population: Data was not collected
Arm/Group | HAI With FOLFOX
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | HAI With FOLFOX
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The study has been terminated due to the Investigator no longer employed at the site and has no access to the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes